CLINICAL TRIAL: NCT05301842
Title: A Phase III, Randomized, Open-Label, Sponsor-Blinded, Multicenter Study of Durvalumab in Combination With Tremelimumab ± Lenvatinib Given Concurrently With TACE Compared to TACE Alone in Patients With Locoregional Hepatocellular Carcinoma (EMERALD-3)
Brief Title: Evaluate Durvalumab and Tremelimumab +/- Lenvatinib in Combination With TACE in Patients With Locoregional HCC
Acronym: EMERALD-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D910VC00001; 2023-508701-24-00 (Registry Identifier: CITS (EU)); 2021-003822-54 (EudraCT Number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Locoregional HCC; Durvalumab; Tremelimumab; Lenvatinib; TACE; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — tremelimumab; durvalumab; lenvatinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Tremelimumab, Durvalumab and Lenvatinib in combination with Transarterial Chemoembolization (TACE)
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Procedure: Transarterial Chemoembolization (TACE); Drug: Lenvatinib
- Arm B (Experimental): Tremelimumab and Durvalumab in combination with Transarterial Chemoemobolization (TACE)
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Procedure: Transarterial Chemoembolization (TACE)
- Arm C (Active Comparator): Transarterial Chemoembolization (TACE)
  Interventions: Procedure: Transarterial Chemoembolization (TACE)

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab IV (intravenous)
  Other Names: MEDI1123
  Arms: Arm A; Arm B
Drug: Durvalumab — Durvalumab IV (intravenous)
  Other Names: MEDI4736
  Arms: Arm A; Arm B
Procedure: Transarterial Chemoembolization (TACE) — TACE (chemo and embolic agent injection into the hepatic artery)
  Other Names: DEB-TACE and cTACE
Drug: Lenvatinib — Lenvatinib (oral)
  Other Names: Lenvima
  Arms: Arm A

SUMMARY:
A global study to evaluate transarterial chemoembolization (TACE) in combination with durvalumab, tremelimumab and lenvatinib therapy in patients with locoregional hepatocellular carcinoma

DETAILED DESCRIPTION:
This is a Phase III, parallel, randomized, open-label, sponsor-blinded, 3-arm, multicenter, international study assessing the efficacy and safety of durvalumab + tremelimumab + TACE with or without lenvatinib compared with TACE alone in participants with locoregional HCC not amenable to curative therapy (eg, surgical resection, transplantation, or ablation).

ELIGIBILITY:
Inclusion Criteria:

* No evidence of extrahepatic disease
* Disease not amenable to curative surgery or transplantation or curative ablation but disease amenable to TACE
* Child Pugh score class A
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* Measurable disease by Modified Response Criteria in Solid Tumors (mRECIST) criteria
* Adequate organ and marrow function

Exclusion Criteria:

* History of symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardia arrhythmia
* History of hepatic encephalopathy
* Major portal vein thrombosis visible on baseline imaging
* Uncontrolled arterial hypertension
* Co-infection with HBV and HDV

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) for Arm A vs Arm C | Approximately 5 years
  PFS is defined as time from randomization until progression per RECIST 1.1 as assessed by BICR or death due to any cause

SECONDARY OUTCOMES:
Overall Survival (OS) for Arm A vs Arm C | Approximately 5 years
  OS is defined as the time from the date of randomization until death due to any cause
Progression Free Survival (PFS) for Arm B vs Arm C | Approximately 5 years
  PFS is defined as time from randomization until progression per RECIST 1.1 as assessed by BICR or death due to any cause
Overall Survival (OS) for Arm B vs Arm C | Approximately 5 years
  OS is defined as the time from the date of randomization until death due to any cause

CONTACTS AND LOCATIONS:
Locations (151):
- United States (12):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Yuma, Arizona
  - Research Site, Glendale, California
  - Research Site, Atlanta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Santa Fe, New Mexico
  - Research Site, Commack, New York
  - Research Site, New York, New York
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Ghent
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Brasília
  - Research Site, Niterói
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (24):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Lanzhou
  - Research Site, Lishui
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Neijiang
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- Egypt (3):
  - Research Site, Al Mansurah
  - Research Site, Cairo
  - Research Site, Shebeen El Kom
- France (10):
  - Research Site, Angers
  - Research Site, Clichy
  - Research Site, Créteil
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (13):
  - Research Site, Bonn
  - Research Site, Chemnitz
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Ulm
- India (8):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, New Delhi
- Italy (6):
  - Research Site, Arezzo
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Tricase
- Japan (18):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kashihara-shi
  - Research Site, Kashiwa
  - Research Site, Kumamoto
  - Research Site, Mitaka-shi
  - Research Site, Morioka
  - Research Site, Musashino-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Tokushima
  - Research Site, Tsu
  - Research Site, Yokohama
- Malaysia (5):
  - Research Site, Bandar Puncak Alam
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Mexico (4):
  - Research Site, Guadalajara, Jalisco
  - Research Site, México
  - Research Site, San Luis Potosí City
  - Research Site, Tuxtla Gutiérrez
- Philippines (5):
  - Research Site, Davao City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Vila Real
- Puerto Rico (2):
  - Research Site, Hato Rey Central
  - Research Site, San Juan
- Saudi Arabia (2):
  - Research Site, Jeddah
  - Research Site, Riyadh
- South Korea (5):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Junggu
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Donostia / San Sebastian
  - Research Site, Madrid
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home